CLINICAL TRIAL: NCT02709005
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter Trial to Assess the Safety and Efficacy of 5% Monolaurin Vaginal Gel Administered Intravaginally for the Treatment of Bacterial Vaginosis
Brief Title: Safety and Efficacy of 5% Monolaurin Vaginal Gel Administered Intravaginally for the Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0021; HHSN272201300017I
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2017-07-19

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Vaginosis; Monolaurin Vaginal Gel
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5% Monolaurin Vaginal Gel (Experimental): 80 subjects will receive 5% Monolaurin Gel twice daily for three successive days for a total of 6 doses
  Interventions: Drug: 5% Monolaurin Vaginal Gel
- Vehicle Placebo (Placebo Comparator): 40 subjects will receive placebo Gel twice daily for three successive days for a total of 6 doses
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 5% Monolaurin Vaginal Gel — Monolaurin Vaginal Gel is a clear and colorless, non-sterile glycol-based gel for vaginal administration , and commonly referred to as glycerol monolaurate (GML). Each subject will receive intravaginal gel twice daily for three successive days for a total of 6 doses. There will be 3 clinic visits over 30 days.
  Arms: 5% Monolaurin Vaginal Gel
Other: Placebo — The placebo gel is a clear to opaque, colorless to light gray, non-sterile glycol-based gel for vaginal administration. The placebo gel contains the same excipients as the Monolaurin vaginal gel. Each subject will receive intravaginal gel twice daily for three successive days for a total of 6 doses. There will be 3 clinic visits over 30 days.
  Arms: Vehicle Placebo

SUMMARY:
This is a Phase II, Double-Blind, Randomized, Placebo-Controlled, Multi-center Trial enrolling 120 subjects with Bacterial Vaginosis who will be randomized at a ratio of 2:1 to receive active test article (5% Monolaurin Vaginal Gel) or placebo (vehicle). The primary objective is to assess the safety and tolerability of 5% Monolaurin Vaginal Gel compared to vehicle placebo gel (excipients only) and to assess the efficacy by clinical cure rate of 5% Monolaurin Vaginal Gel compared to vehicle placebo gel at Visit 2.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is a disease of the vagina caused by bacteria. The most common symptom of BV is an abnormal homogeneous off-white vaginal discharge (especially after sex) with an unpleasant smell. This is a Phase II, Double-Blind, Randomized, Placebo-Controlled, Multi-center Trial enrolling 120 women, 18-50 years old, with clinical evidence of bacterial vaginosis. Subjects will be randomized at a ratio of 2:1 to receive active test article (5% Monolaurin Vaginal Gel) or placebo (vehicle) as outpatient therapy. Subjects will be stratified by first time episode of bacterial vaginosis or recurrent bacterial vaginosis. The primary objectives of this study are: 1) To assess the safety and tolerability of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel (excipients only) and 2) To assess the efficacy by clinical cure rate of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel at Visit 2. The secondary objectives are : 1) To evaluate the therapeutic cure rate of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel at Visits 2 and 3, 2) To evaluate the clinical cure rate of 5% Monolaurin Vaginal Gel compared to Vehicle Placebo Gel at Visit 3, 3) To evaluate the changes in Nugent's criteria of vaginal bacterial flora at Visits 2 and 3. This study is expected to last for 13 months, with subject participation duration being 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-breastfeeding females between the ages of 18 and 50 years, inclusive
* Women of childbearing potential* must agree to practice reliable contraception** for the 28-day period before enrollment through 30 days following treatment.

  *(not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy, or who have not been postmenopausal for >/=1 year)

  ** Acceptable birth control methods for the purposes of this study may include, but are not limited to, abstinence from intercourse with a male partner, monogamous relationship with vasectomized partner, barrier methods to include condoms and diaphragms, intrauterine devices, and licensed hormonal methods. NuvaRing® contraceptive use will be prohibited from this study since the device can alter vaginal secretions
* Presenting with signs of BV (as per Amsel Criteria). Subjects must meet any three of the four criteria for enrollment*

  *Presence of discharge, greater than or equal to 20% clue cells on wet prep, positive "whiff test" on KOH prep, vaginal pH of greater than 4.5
* Not currently menstruating or expected to in the next 4 days
* Able to understand and comply with planned study procedures
* Willing to abstain from sexual intercourse, insertion of tampons, douches, or other intravaginal medications or objects between Visit 1 and Visit 2 and 48 hours prior to Visit 3
* Provide written informed consent before initiation of any study procedures and be available for all study visits
* No known history of HIV

Exclusion Criteria:

-Signs or symptoms of vaginal/cervical/pelvic infection on screening or clinical diagnosis of vaginal/cervical/pelvic infection in the past 14 days.

* (including but not limited to yeast vulvovaginitis, chlamydia, gonorrhea, trichomonas, genital ulcer disease, pelvic inflammatory disease). Self-treatment for presumed yeast vaginitis is not an exclusion if treatment was discontinued 7 days or greater prior to enrollment

  * Treatment for BV within the past 14 days
  * Cervical or vaginal high grade squamous intraepithelial dysplasia (HSIL), atypical glandular cells of uncertain significance (AGUS) or cervical intraepithelial neoplasia grade 2 (CIN2) or higher*
* Atypical squamous cells of undetermined significance (ASCUS), low grade squamous intraepithelial lesion (LSIL) or cervical intraepithelial neoplasia grade 1 (CIN1) are acceptable. Individuals with a history of atypical glandular cells of uncertain significance (AGUS), HSIL or CIN2 and who have received subsequent evaluation and/or treatment with follow up normal PAP smear are eligible. Patient report will be accepted

  * History of undiagnosed vaginal bleeding
  * Use of a systemic, vaginal, or perineal antibiotic within 7 days prior to enrollment in this study
  * Use of an immunosuppressive or immunomodulatory drug* for two or more consecutive weeks within 6 months prior to enrollment
* such as >0.5 mg/kg/day or >/=20 mg total dose/day of prednisone orally or >800 µg of inhaled beclomethasone (nasal and non-genital topical steroids are allowed)

  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to Monolaurin Vaginal Gel
  * Uncontrolled concurrent illness*. Subjects with a history of organ or marrow transplant are excluded.
* Including, but not limited to, ongoing or active infection, active liver, kidney or autoimmune diseases (a history of thyroid disease will be permitted as long as the thyroid disease is now stable), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

  * Acute illness within 3 days before receipt of study product (per investigator's discretion)
  * Pregnant women and women who are planning to become pregnant within 30 days after the final study dose, or women who are breastfeeding
  * Immunosuppression as a result of an underlying illness or treatment or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months
  * Active neoplastic disease* or a history of any hematologic malignancy. Active neoplastic disease is defined as neoplastic disease or treatment for neoplastic disease within the past 5 years
* (excluding non-melanoma skin cancer)

  -Received an experimental agent* within 30 days before receipt of study product or expect to receive an experimental agent during the 1 month study period.
* (vaccine, drug, biologic, device, blood product, or medication)

  * Any condition that would place the subject at an unacceptable risk of injury, render her unable to meet the requirements of the protocol, or that may interfere with successful completion of the study
  * A history of alcohol or drug abuse* during the previous 1 year that in the opinion of the site investigator would interfere with study procedures
* For example, daily excessive alcohol use or frequent binge drinking as determined by the investigator, or daily marijuana use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Duke Human Vaccine Institute - Duke Clinical Vaccine Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women, 18-50 years old, with clinical evidence of bacterial vaginosis, were identified during a routine clinic visit, referred by their care provider, or recruited directly to the research clinic between May 11, 2016 and November 16, 2017.
Groups:
- 5% Monolaurin Vaginal Gel: Monolaurin Vaginal Gel is a clear and colorless, non-sterile glycol-based gel for vaginal administration, and commonly referred to as glycerol monolaurate (GML). Participants were to receive intravaginal gel twice daily for three successive days for a total of 6 doses.
- Vehicle Placebo: The placebo gel is a clear to opaque, colorless to light gray, non-sterile glycol-based gel for vaginal administration. The placebo gel contains the same excipients as the Monolaurin vaginal gel. Participants were to receive intravaginal gel twice daily for three successive days for a total of 6 doses.
Period: Overall Study
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Started | 73 | 36
Completed | 69 | 35
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo | Total
Number analyzed (Participants) | 73 | 36 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 36 | 109
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (8.4) | 31.3 (8.4) | 30.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 36 | 109
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 68 | 31 | 99
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 45 | 19 | 64
  White | 26 | 11 | 37
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 36 | 109
Nugent score <4 [Count of Participants; unit: Participants] — A vaginal swab for bacteriological assessment of BV by Nugent criteria was performed. The Nugent score utilizes a 10-point scale for evaluation of vaginal flora. The Nugent score can range from 0 to 10. A score of 7 to 10 is consistent with BV while 4-6 is considered intermediate and 0-3 is negative for BV.
  Participants | 7 | 2 | 9
Positive HIV, Chlamydia, or Neisseria gonorrhoeae test [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cure in Each Study Arm
Description: A clinical cure was defined by normal Amsel criteria, including: normal physiological vaginal discharge, whiff test negative for any amine "fishy" odor, saline wet mount less than 20% for clue cells, and vaginal pH is <=4.5. All four criteria had to be normal with none of the clinical failure criteria met to be considered a clinical cure. A clinical failure was defined by at least one of the following: one or more abnormal Amsel criteria, early discontinuation of study therapy due to lack of treatment effect, use of any vaginosis therapy other than study product during the study, or in the investigator's opinion, required additional treatment for vaginosis.
Time Frame: Visit 2 (Day 8-15)
Population: The mITT population includes randomized participants who met inclusion/exclusion criteria, excluding those with Nugent score <4 at Visit 1 or a positive Visit 1 HIV, Chlamydia, or Neisseria gonorrhoeae test. In the event of an error in randomization or study product administration, participants were grouped by their intended randomized assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 64 | 32
Participants | 11 | 8
Statistical Analysis 1: Comparison: 5% Monolaurin Vaginal Gel vs Vehicle Placebo; The null hypothesis was that there was no difference in participants with clinical cure between study arms, with a two-sided alternative considering the possibility of a difference in either direction. The statistical informational goal for the study of 90 participants eligible in the modified Intent-to-Treat (mITT) efficacy population was an ad-hoc sample size determined by logistical considerations, as there was insufficient pilot data upon which to base more formal sample size calculations; Test type: Superiority; p = 0.420, Fisher Exact — The test was conducted using a Fisher's exact test at the 5% two-sided level of significance level without adjustment for multiplicity; Risk Difference (RD) = -0.08, 95% CI 2-sided [-0.26 to 0.08] — Difference in Proportion of Participants with Clinical Cure between 5% Monolaurin Vaginal Gel and Placebo Gel

2. Primary Outcome: Number of Participants Reporting Solicited Urogenital Adverse Events (AEs) Following the First Dose of the Study Product
Description: Solicited event assessments were captured on a memory aid starting on Day 1, the first day of therapy and continuing for 5 days. The participant recorded the presence and intensity of vulvovaginal solicited events on the memory aid. Any symptom that was present at the time that the participant was screened was considered as baseline and not reported as a solicited urogenital AE. However, if the symptom deteriorated during the reporting period, it was considered an AE. If a symptom was reported that was not present at baseline, it too was considered an AE. Any symptoms still present on Day 5 were followed by participant memory aid notations until symptom resolution. Solicited events collected include vaginal odor, vaginal pain, vaginal tenderness, vaginal itching, vaginal dryness, vaginal discharge, and vaginal inflammation. Severity of solicited events symptoms were graded as mild, moderate, or severe according to the grading table in the protocol.
Time Frame: Days 1 through 5
Population: The safety population includes all randomized participants who received at least one dose of study treatment. If a subject did not have solicited symptom data she was not included. In the event of an error in randomization or study product administration (i.e., incorrect product), participants were grouped by the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 71 | 37
Participants
  Any Symptom | 50 | 21
  Vaginal Odor | 10 | 6
  Vaginal Pain | 16 | 5
  Vaginal Tenderness | 10 | 2
  Vulvar/Vaginal Itching | 23 | 9
  Vaginal Dryness | 10 | 3
  Vaginal Discharge | 12 | 8
  Vulvar Inflammation | 9 | 2
Statistical Analysis 1: Comparison: 5% Monolaurin Vaginal Gel vs Vehicle Placebo; The null hypothesis was that there was no difference in participants with solicited urogenital AEs between study arms, with a two-sided alternative considering the possibility of a difference in either direction; Test type: Superiority; p = 0.200, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.14, 95% CI 2-sided [-0.06 to 0.33] — Difference in Proportion of Participants Experiencing Solicited Events between 5% Monolaurin Vaginal Gel and Placebo Gel

3. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Considered Product-related
Description: The number of participants in each treatment group with product-related SAEs was assessed. An AE was considered "serious" if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, or a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalizations could be considered serious when, based upon appropriate medical judgment, they could jeopardize the participant and require medical or surgical intervention to prevent one of the outcomes listed. An AE was considered related if there was a reasonable possibility that the study product caused the AE, meaning that there is evidence to suggest a causal relationship between the study product and the AE.
Time Frame: Visit 1 (Day 1) through Visit 3 (Day 22-31)
Population: The safety population includes all randomized participants who received at least one dose of study treatment. In the event of an error in randomization or study product administration (i.e., incorrect product), participants were grouped by the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 72 | 37
Participants | 0 | 0
Statistical Analysis 1: Comparison: 5% Monolaurin Vaginal Gel vs Vehicle Placebo; The null hypothesis was that there was no difference in participants with related SAEs between study arms, with a two-sided alternative considering the possibility of a difference in either direction; Test type: Superiority; No SAEs were reported; therefore the Fisher's Exact Test was not performed; Risk Difference (RD) = 0

4. Secondary Outcome: Number of Participants With Therapeutic Cure in Each Study Arm
Description: Therapeutic cure was defined as both a clinical cure and a bacteriological cure. All four Amsel criteria had to be normal with none of the clinical failure criteria listed met to be considered a clinical cure, including normal physiological vaginal discharge, whiff test negative for any amine "fishy" odor, saline wet mount less than 20% for clue cells, and vaginal pH is <=4.5. A clinical failure was defined by at least one of the following: one or more abnormal Amsel criteria, early discontinuation of study therapy due to lack of treatment effect, use of any vaginosis therapy other than study product during the study, or in the investigator's opinion, required additional treatment for vaginosis. A vaginal swab for bacteriological assessment of BV by Nugent criteria was performed. The Nugent score can range from 0 to 10. Bacteriological cure of BV was defined as a normal Nugent score of 0-3. Participants who were clinical failures, or had a Nugent score >3 were therapeutic failures.
Time Frame: Visit 2 (Day 8-15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 64 | 32
Participants | 2 | 1
Statistical Analysis 1: Comparison: 5% Monolaurin Vaginal Gel vs Vehicle Placebo; The null hypothesis was that there was no difference in participants with therapeutic cure between study arms, with a two-sided alternative considering the possibility of a difference in either direction; Test type: Superiority; p > 0.999, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.13 to 0.08] — Difference in Proportion of Participants with Therapeutic Cure between 5% Monolaurin Vaginal Gel and Placebo Gel

5. Secondary Outcome: Number of Participants With Therapeutic Cure in Each Study Arm
Description: as for outcome 4
Time Frame: Visit 3 (Day 22-31)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 64 | 32
Participants | 0 | 3
Statistical Analysis 1: Comparison: 5% Monolaurin Vaginal Gel vs Vehicle Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.035, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.09, 95% CI 2-sided [-0.24 to -0.01] — Difference in Proportion of Participants with Therapeutic Cure between 5% Monolaurin Vaginal Gel and Placebo Gel

6. Secondary Outcome: Number of Participants With Nugent Score of 3 or Less (Negative for BV) in Each Study Arm
Description: A vaginal swab for bacteriological assessment of BV by Nugent criteria was performed. The Nugent score utilizes a 10-point scale for evaluation of vaginal flora. The Nugent score can range from 0 to 10. A score of 7 to 10 is consistent with BV while 4-6 is considered intermediate and 0-3 is negative for BV. Bacteriological cure of BV was defined as a normal Nugent score of 0-3.
Time Frame: Visit 2 (Day 8-15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 61 | 31
Participants | 2 | 1

7. Secondary Outcome: Number of Participants With Nugent Score of 3 or Less (Negative for BV) in Each Study Arm
Description: as for outcome 6
Time Frame: Visit 3 (Day 22-31)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 60 | 31
Participants | 5 | 8

8. Secondary Outcome: Number of Participants With Nugent Score of 4-6 (Intermediate BV) in Each Study Arm
Description: as for outcome 6
Time Frame: Visit 2 (Day 8-15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 61 | 31
Participants | 8 | 3

9. Secondary Outcome: Number of Participants With Nugent Score of 4-6 (Intermediate BV) in Each Study Arm
Description: as for outcome 6
Time Frame: Visit 3 (Day 22-31)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 60 | 31
Participants | 9 | 3

10. Secondary Outcome: Number of Participants With Clinical Cure in Each Study Arm
Description: A clinical cure was defined by normal Amsel criteria, including: normal physiological vaginal discharge, whiff test negative for any amine "fishy" odor, saline wet mount less than 20% for clue cells, and vaginal pH is <=4.5. All four criteria had to be normal with none of the clinical failure criteria met to be considered a clinical cure. A clinical failure was defined by at least one of the following: one or more abnormal Amsel criteria, early discontinuation of study therapy due to lack of treatment effect, use of any vaginosis therapy other than study product during the study, or in the investigator's opinion, requires additional treatment for vaginosis. Participants who did not have enough information to determine a clinical cure or clinical failure status were not evaluable for clinical cure.
Time Frame: Visit 3 (Day 22-31)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 64 | 32
Participants | 10 | 5
Statistical Analysis 1: Comparison: 5% Monolaurin Vaginal Gel vs Vehicle Placebo; The null hypothesis was that there was no difference in participants with clinical cure between study arms, with a two-sided alternative considering the possibility of a difference in either direction; Test type: Superiority; p > 0.999, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.18 to 0.14] — Difference in Proportion of Participants with Clinical Cure between 5% Monolaurin Vaginal Gel and Placebo Gel

11. Secondary Outcome: Number of Participants Experiencing Non-laboratory Non-solicited AEs Following the First Dose of the Study Product
Description: The number of participants who experienced non-laboratory, non-solicited AEs following the first dose of the study product through Visit 3 (Day 22-31) was assessed. Events involving laboratory parameters that were not collected as part of the protocol were counted as non-laboratory, non-solicited adverse events.
Time Frame: Visit 1 (Day 1) through Visit 3 (Day 22-31)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 72 | 37
Participants | 52 | 20

12. Secondary Outcome: Number of Participants Experiencing Laboratory AEs Following the First Dose of the Study Product
Description: The number of participants experiencing laboratory AEs following the first dose of the study product was assessed at Visit 2 (Day 8-15). A laboratory abnormality was considered an adverse event if there was a worsening of the laboratory value at Visit 2 from the baseline value and it increased in laboratory toxicity grading from the baseline toxicity grading. Protocol-defined hematology parameters assessed were white blood cells, hemoglobin, platelets, and neutrophils. Protocol-defined clinical chemistry parameters assessed were creatinine, AST, ALT, total bilirubin, and glucose (random).
Time Frame: Visit 2 (Day 8-15)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
Number analyzed (Participants) | 72 | 37
Participants
  Any Laboratory AE | 12 | 7
  Hemoglobin decrease | 2 | 4
  White blood cells Increase | 3 | 0
  White blood cells Decrease | 1 | 0
  Platelets Decrease | 1 | 0
  Neutrophils Decrease | 2 | 0
  Glucose Decrease | 1 | 0
  Glucose Increase | 0 | 1
  Creatinine Increase | 1 | 1
  AST Increase | 1 | 0
  ALT Increase | 1 | 2
  Bilirubin Increase | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited urogenital AEs were collected following the first dose of the study product (Day 1) through Day 5. Laboratory AEs were collected at Visit 2 (Day 8-15). Serious adverse events and non-laboratory non-solicited AEs were collected following the first dose of the study product (Day 1) through Visit 3 (Day 22-31).
Description: Solicited symptoms were counted as AEs if they developed or worsened after the baseline symptom toxicity. Laboratory abnormalities for protocol-specified labs were considered AEs if they worsened at Visit 2 from the baseline value and increased in laboratory toxicity grading from the baseline toxicity grading. Protocol-defined laboratory parameters collected were white blood cells, hemoglobin, platelets, neutrophils, creatinine, AST, ALT, total bilirubin, and glucose (random).
Arm/Group | 5% Monolaurin Vaginal Gel | Vehicle Placebo
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/37
Other Adverse Events (participants affected / at risk) | 59/72 | 28/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5% Monolaurin Vaginal Gel (N=72) | Vehicle Placebo (N=37)
Vaginal Odour (Reproductive system and breast disorders) | 10/71 (10) | 6 (6) — Solicited on the memory aid for 5 days after first dose of product and reviewed in the clinic at Visit 2 (Day 8-15)
Vulvovaginal Pain (Reproductive system and breast disorders) | 22/71 (22) | 5 (5) — Solicited on the memory aid for 5 days after first dose of product and reviewed in the clinic at Visit 2 (Day 8-15)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 23/71 (23) | 9 (9) — Solicited on the memory aid for 5 days after first dose of product and reviewed in the clinic at Visit 2 (Day 8-15)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 10/71 (10) | 3 (3) — Solicited on the memory aid for 5 days after first dose of product and reviewed in the clinic at Visit 2 (Day 8-15)
Vaginal Discharge (Reproductive system and breast disorders) | 12/71 (12) | 8 (8) — Solicited on the memory aid for 5 days after first dose of product and reviewed in the clinic at Visit 2 (Day 8-15)
Vulvovaginal Inflammation (Reproductive system and breast disorders) | 9/71 (9) | 2 (2) — Solicited on the memory aid for 5 days after first dose of product and reviewed in the clinic at Visit 2 (Day 8-15)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 5 (5)
Vulvovaginal Mycotic Infection (Infections and infestations) | 6 (7) | 3 (3)
Vaginal Odour (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 30 (46) | 4 (6)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) — Protocol-defined blood chemistry tests were performed on Visit 2 samples (Day 8-15)
Haemoglobin decreased (Investigations) | 2 (2) | 4 (4) — Protocol-defined hematology tests were performed on Visit 2 samples (Day 8-15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT02709005/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02709005/SAP_001.pdf